CLINICAL TRIAL: NCT03822065
Title: A Randomized, Open-Label, 2-Period, Crossover Trial to Assess the Relative Bioavailability of 80 mg LY03005 After Single Dose Administration to Healthy Subjects Under Fed Versus Fasted Conditions
Brief Title: A Relative Bioavailability Food Effect Study of LY03005
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LY03005/CT-USA-105
Record Dates: First submitted 2019-01-25; First posted 2019-01-30 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-01

CONDITIONS: Major Depressive Disorder
Keywords: Depressive Disorder, Major; Depressive Disorder; Mood Disorders; Mental Disorders; Desvenlafaxine Succinate; Serotonin and Noradrenaline Reuptake Inhibitors; Neurotransmitter Uptake Inhibitors; Membrane Transport Modulators; Molecular Mechanisms of Pharmacological Action; Neurotransmitter Agents; Physiological Effects of Drugs; Antidepressive Agents; Psychotropic Drugs
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder; Mood Disorders; Mental Disorders | interventions — Desvenlafaxine Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence 1: LY03005 Fed Crossover to Fasted (Experimental): Sequence 1 will receive a single oral dose of LY03005 (80 mg) under fed conditions in Treatment Period 1 and a single oral dose of LY03005 (80 mg) under fasted conditions in Treatment Period 2.
  Interventions: Drug: LY03005
- Sequence 2: LY03005 Fasted Crossover to Fed (Experimental): Sequence 2 will receive a single oral dose of LY03005 (80 mg) under fasted conditions in Treatment Period 1 and a single oral dose of LY03005 (80 mg) under fed conditions in Treatment Period 2.
  Interventions: Drug: LY03005

INTERVENTIONS:
Drug: LY03005 — 80 mg oral tablet single dose
  Other Names: Desvenlafaxine

SUMMARY:
The objective if this study is to assess the relative bio-availability of single oral doses of 80 mg LY03005 tablets administered to healthy subjects under fed versus fasted conditions in a 2-period, crossover trial.

DETAILED DESCRIPTION:
Thirty-two (32) eligible healthy subjects between ages of 18-50 years old will be enrolled and randomized to either Sequence 1 (fed to fasted state) versus Sequence 2 (fasted to fed state) at a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving informed consent and complying with trial procedures;
2. Male and female subjects between the ages of 18 and 50 years, inclusive;
3. Considered healthy by the Investigator based on a detailed medical history, full physical examination, clinical laboratory tests, 12-lead ECG, and vital signs;
4. Nonsmoker, defined as not having smoked or used any form of tobacco for at least 6 months before Screening based on subject report;
5. Body mass index (BMI) of 19 to 30 kg/m2 inclusive and body weight >/= 50 kg;
6. Willing and able to adhere to trial procedures and to be confined at the clinical research unit (CRU).
7. All female subjects (childbearing potential and non-childbearing potential) must have a negative serum pregnancy test result at Screening. In addition, female subjects must meet 1 of the following 3 conditions: (a) postmenopausal for at least 12 months without an alternative medical cause, (ii) surgically sterile (hysterectomy, bilateral oophorectomy, bilateral salpingectomy, or bilateral tubal occlusion) based on subject report, or (iii) if of childbearing potential and heterosexually active, practicing or agree to practice a highly effective method of contraception. Highly effective methods of birth control include an intrauterine device (IUD), intrauterine hormone-releasing system (IUS), and contraceptives (oral, skin patches, or implanted or injectable products) using combined or progestogen-only hormonal contraception associated with inhibition of ovulation. A vasectomized male partner is an acceptable birth control method if the vasectomized partner is the sole sexual partner of the female subject and the vasectomized partner has received medical confirmation of surgical success. Highly effective methods of birth control must be used for at least 14 days prior to study drug dosing, through the end of study (EOS) visit or early termination, and for a minimum of 1 month after the last dose of study drug to minimize the risk of pregnancy. Sexually active, fertile, male subjects must be willing to use acceptable contraception methods (such as double-barrier methods of a combination of male condom with either cap, diaphragm, or sponge with spermicide) from the first dose of study drug through the EOS visit or early termination, and for a minimum of 1 month after the last dose of study drug.

Exclusion Criteria:

1. Clinically significant past medical history of gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematologic, psychiatric (including life-long history of depression and/or anxiety), renal, hepatic, bronchopulmonary, neurologic, immunologic, ophthalmological, or lipid metabolism disorders; or drug hypersensitivity; or any condition that in the judgement of the Investigator will affect the trial results or the subject's safety;
2. History of suicide attempt in the past 12 months and/or seen by the Investigator as having a significant history of risk of suicide or homicide;
3. History or presence of malignancy other than adequately treated and cured basal cell skin cancer, squamous cell skin cancer, or in-situ cervical cancer, within 5 years prior to screening;
4. Clinically relevant illness within 1 month prior to Screening or at Screening that may interfere with the conduct of this trial;
5. Medically uncontrolled high blood pressure with mean systolic blood pressure >140 mmHg or mean diastolic blood pressure >90 mmHg at Screening after 3 measurements (after at least 5 minutes of rest in a seated position);
6. History of Long QT Syndrome (LQTS) or a marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms);
7. Positive blood screen for HIV, hepatitis B surface antigen (HBsAg), or hepatitis C antibody;
8. History of seizure (history of febrile seizure allowed);
9. Hospital admission or major surgery within 30 days prior to Screening;
10. Participation in any other investigational drug trial within 30 days prior to Screening;
11. History of prescription drug abuse or illicit drug use within 6 months prior to Screening;
12. History of alcohol abuse according to medical history within 6 months prior to Screening;
13. Positive screen for alcohol and/or drugs of abuse;
14. Tobacco use within 6 months prior to Screening based on subject report or positive nicotine screen;
15. History of intolerance or hypersensitivity to ODV or medicines containing ODV or its precursor venlafaxine;
16. Participation in a previous clinical trial of either LY03005 or ODV or medicines containing ODV or its precursor, venlafaxine, within 30 days prior to Screening;
17. Unwillingness or inability to comply with food and beverage restrictions during trial participation;
18. Donation of blood of more than 1 unit (approximate 450 mL) or blood products or acute loss of blood during the 90 days prior to Screening;
19. Use of prescription or over-the-counter (OTC) medications and herbals (including St John's Wort, herbal teas, garlic extracts) within 14 days prior to dosing (Note: Use of acetaminophen at <3g/day is permitted until 24 hours prior to dosing).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2019-02-16 (Actual); Study Completion 2019-02-16 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Parameters | PK samples drawn at predose (within 30 minutes prior to dosing) and at 1, 2, 3, 4 (±5 minutes), 6, 8, 10, 12, 16, 24, 32, 48, and 72 hours (±15 minutes) after the dose.
  Area under the concentration-time curve (AUC)
Pharmacokinetic Parameters | PK samples drawn at predose (within 30 minutes prior to dosing) and at 1, 2, 3, 4 (±5 minutes), 6, 8, 10, 12, 16, 24, 32, 48, and 72 hours (±15 minutes) after the dose.
  Maximum concentration (Cmax) for the Pharmacokinetics (PK) of O-desmethyl-venlafaxine (ODV) from LY03005

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Booth, MD, DVM, Study Director — Luye Pharma.
Locations (1):
- Pharmaron CPC, Inc., Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Drug information — https://druginfo.nlm.nih.gov/drugportal/
- See also: Desvenlafaxine — https://druginfo.nlm.nih.gov/drugportal/name/Desvenlafaxine
- See also: Desvenlafaxine Succinate — https://druginfo.nlm.nih.gov/drugportal/name/desvenlafaxine%20succinate
- See also: U.S. FDA Resources — https://clinicaltrials.gov/ct2/info/fdalinks